CLINICAL TRIAL: NCT06012981
Title: Psychological Treatment in Psychiatric Inpatient Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unforeseen difficulties in recruiting participants.
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Marten Tyrberg, Principal Investigator, Uppsala University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 280468
Record Dates: First submitted 2023-04-28; First posted 2023-08-28 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Compulsory Psychiatric Care Act; Psychosis; Acceptance & Commitment Therapy; Psychiatric Hospitalization; Psychiatric Disorder
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Single-case experimental design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance & Commitment Therapy (ACT) (Experimental): Psyhotherapy based on principles of functional analysis, behavioral activation, and experiential avoidance.
  Interventions: Behavioral: ACT

INTERVENTIONS:
Behavioral: ACT — The treatment is based on a variant of CBT, as briefly referred to before, ACT. In short, the treatment consists of identifying central and important areas of life, and how to approach these even though you are also struggling with persistent and challenging problems. In this study, the treatment intervention is flexibly constructed, focusing on several central principles based on ACT. These can be applied during one or numerous sessions.
  The intervention is a flexible application of clinical functional analysis, as well as a couple of selected interventions which, in terms of experience and in previous studies, have been shown to work well for the current group (24-hour psychiatric patients with complex problems) and which are individually adaptable to the nature of the problem and degree.

SUMMARY:
This study aims to investigate the effect of a brief psychotherapeutic treatment intervention based on ACT, aimed specifically at the vulnerable group of patients in psychiatric 24-hour care treated according to LPT. The study aims to investigate whether a brief number of therapeutic sessions according to ACT during inpatient care produce positive effects on personally relevant life areas for a diagnostically mixed group of patients in a psychiatric intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older.
* Treated according to the compulsory psychiatric care act.
* Meet the criterion of informed consent.

Exclusion Criteria:

* Lack the cognitive ability to acquire the treatment intervention, such as impaired attention, memory, logic and reasoning, and also auditory and visual processing. This will be based on a clinical assessment by the ward team, including the attending psychiatrist and a clinical psychologist.
* Ongoing psychological treatment parallel to the admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Change in Personal Questionnaire | Four times daily, from point of inclusion to after a minimum of five data points (approximately a day and a half) after last treatment session
  Scores range from 1-4 per item (number of items might differ between patients as the measure is individually constructed. Higher scores correspond to worse outcome.
Change in Bull's Eye Values Survey | Four times daily, from point of inclusion to after a minimum of five data points (approximately a day and a half) after last treatment session
  The score ranges from 0-28, higher scores corresponding to better outcome.
Change in PHQ-9 | Four times daily, from point of inclusion to after a minimum of five data points (approximately a day and a half) after last treatment session
  The score ranges from 0-27, higher scores corresponding to worse outcome.
Change in GAD-7 | Four times daily, from point of inclusion to after a minimum of five data points (approximately a day and a half) after last treatment session
  The score ranges from 0-21, higher scores corresponding to worse outcome.
Change in Psy-flex | Four times daily, from point of inclusion to after a minimum of five data points (approximately a day and a half) after last treatment session
  The score ranges from 6-30, higher scores corresponding to better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kent Nilsson, Professor, Study Director — Uppsala University
Locations (1):
- Hospital of Västmanland, Västerås, Västerås, Västmanland County, Sweden

IPD SHARING:
Plan to Share IPD: No